CLINICAL TRIAL: NCT05178693
Title: The Epigenetic Modification of Somatostatin Receptor-2 to Improve Therapeutic Outcome With Lutathera in Patients With Metastatic Neuroendocrine Tumours.
Brief Title: Lutathera and ASTX727 in Neuroendocrine Tumours
Acronym: LANTana
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS - IC03; 21HH6544 (Other: Imperial College London)
Record Dates: First submitted 2021-12-03; First posted 2022-01-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — decitabine and cedazuridine drug combination; lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: ASTX727; Radiation: Lutathera

INTERVENTIONS:
Drug: ASTX727 — Cedazuridine 100mg + 35mg decitabine
Radiation: Lutathera — Peptide receptor radionuclide therapy (PRRT)
  Other Names: lutetium Lu 177 dotatate

SUMMARY:
Patients entered into the study will receive ASTX727 orally for 5 days, prior to receiving Lutathera treatment on Day 8, to determine whether pre-treatment with ASTX727 results in re-expression of somatostatin receptor-2 in patients with metastatic neuroendocrine tumours. The study will use [68Ga]-DOTA-TATE PET to image epigenetic modification of the receptor locus.

DETAILED DESCRIPTION:
Patients with neuroendocrine tumours (NET) who are found to be eligible will receive up to 4 doses of Lutathera on this trial. All participants will receive ASTX727 orally (cedazuridine 100mg + 35mg decitabine) Days 0-5 prior to receiving Lutathera Day 8 +/- 2days. Each cycle will be repeated every 2 months for 4 cycles unless unacceptable toxicity, progression of disease or withdrawal of patients' consent. Restaging will occur after 2 cycles of Lutathera and at the end of treatment. Patients will be followed 3 monthly until disease progression, death or withdrawal of patients' consent.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Be aged 18 or over at the day of signing consent
3. Histologic or cytologic confirmed diagnosis of neuroendocrine tumour
4. Have archival tissue block available or willing to have fresh tissue biopsy if blocks not available
5. Have disease that can be readily biopsied by ultrasound guidance (n=5)
6. Ki67 < 55% (only patients with well differentiated grade 1-3 NETs will be included in the study as patients with poorly differentiated grade 3 NETs have a prognosis of less than 6 months)
7. Progression or intolerance to first line therapy including somatostatin analogues
8. ECOG Performance status 0 - 2
9. No tumoural uptake on [68Ga]-DOTA-TATE or uptake less than background liver
10. Measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
11. Adequate organ function as outlined in the protocol
12. Women of childbearing potential must be willing to use a highly effective method of contraception as outlined in the protocol for the course of the study through 6 months after the last dose of Investigational Medicinal Product (IMP).

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subjects
13. Sexually active males must agree to use an adequate method of contraception as outlined in the protocol starting with the first dose of IMP through 6 months after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

Exclusion Criteria:

1. Previous treatment with either study medication and/or known hypersensitivity to the study medication
2. Serious concurrent medical illness, including serious active infection
3. History of organ transplant
4. Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
5. Has a known history of active Bacillus Tuberculosis (TB).
6. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
7. Bleeding or thrombotic disorders or subjects at risk for severe haemorrhage
8. Is currently participating and receiving therapy or has participated or is participating in a study of an IMP or used an investigational device within 4 weeks of the first dose of IMP.
9. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Principal Investigator (PI).
11. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through to 6 months after the last dose of IMP.
13. Has received a live vaccine within 30 days of first dose of ASTX727 administration. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
14. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease and stereotactic radiotherapy to the CNS
15. Other clinically significant co-morbidities that could compromise the subject's participating in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
To determine whether pre-treatment with ASTX727 results in re-expression of SSTR2 in patients with metastatic NETs, using [68Ga]-DOTA-TATE to image epigenetic modification of the SSTR2 locus allowing subsequent treatment with Lutathera | Through study completion, an average of 1 year
  This outcome will be assessed using a specific PET scan

SECONDARY OUTCOMES:
To assess tolerability of combination therapy | Through study completion, an average of 1 year
  This outcome will be assessed using CTCAE v5.0
To assess response to treatment using conventional imaging | Through study completion, an average of 1 year
  This outcome will be assessed using standard of care CT scans
To assess patients quality of life during treatment | Through study completion, an average of 1 year
  This will be assessed using standardised quality of life questionnaires, which will be given to the patients
To assess progression free survival | Through study completion, an average of 1 year
  This will be the time until patients show progressive disease on their routine CT scans

CONTACTS AND LOCATIONS:
Overall Officials: Rohini Sharma, Professor, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospital, London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murphy R, Chander G, Martinez M, Ward C, Khan SR, Naik M, Barwick T, Aboagye E, Sharma R. Study protocol of LANTana: a phase Ib study to investigate epigenetic modification of somatostatin receptor-2 with ASTX727 to improve therapeutic outcome with [177Lu]Lu-DOTA-TATE in patients with metastatic neuroendocrine tumours, UK. BMJ Open. 2023 Oct 24;13(10):e075221. doi: 10.1136/bmjopen-2023-075221. PMID 37879695